CLINICAL TRIAL: NCT04429308
Title: PDT Versus the Combination of Jessner's Solution and 35% TCA for Treatment of Actinic Keratoses on Upper Extremities: A Randomized Controlled Split-arm Trial
Brief Title: PDT vs Peels for Treatment of Actinic Keratoses
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00211723
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Chemexfoliation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Photodynamic Therapy (Active Comparator): One upper arm will be exposed to blue light therapy
  Interventions: Procedure: Photodynamic Therapy
- Chemical Peels (Active Comparator): One upper arm will be exposed to Jessner's Solution AND 35% Trichloroacetic acid peel
  Interventions: Drug: Chemical Peels

INTERVENTIONS:
Procedure: Photodynamic Therapy — Photodynamic Therapy consists of (Levulan Kerastick (aminolevulinic acid HCL) topical solution, 20% + BLU-U Photodynamic Light Therapy)
  Other Names: PDT
  Arms: Photodynamic Therapy
Drug: Chemical Peels — Chemical peels consists of a combination of Jessner's Solution: Composed of Salicylic Acid (14%), Medical Grade Lactic Acid (14%), Medical Grade Resorcinol (14%), Denatured Ethyl Alcohol AND 35% Trichloroacetic acid peels
  Arms: Chemical Peels

SUMMARY:
The purpose of this study is to to compare photodynamic therapy (PDT) versus the combination of Jessner's solution and 35% trichloroacetic acid (TCA) chemical peels for the treatment of actinic keratoses on upper extremities.

This is a randomized clinical trial. Approximately 60 participants with actinic keratoses on both upper arms will be randomized to have one arm receive photodynamic therapy, while the contralateral arm receives Jessner's solution followed immediately by 35% TCA. AKs will be counted before treatment and 2-8 weeks after treatment. This study is a pilot study designed to determine the feasibility of this procedure.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Interested in receiving treatment for actinic keratoses on the bilateral upper arms
3. In good general health as assessed by the investigator
4. Participants must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

1. Patient pregnant or nursing
2. Patient with extensive concurrent skin conditions (such as eczema, psoriasis, etc) on upper extremities that would interfere with treatment as determined by the treating physician
3. Subject unwilling to sign an IRB approved consent form
4. Participants who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of total AKs cleared | 2-8 weeks after treatments
  Percentage of total AKs cleared will be calculated by counting the number of AKs before treatment and 2-8 weeks after treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No